CLINICAL TRIAL: NCT04419220
Title: Evaluating Reproducibility of Flow Measurements in the Superior Mesenteric Artery in Healthy Male Subjects Using Doppler Ultrasound
Brief Title: Reproducibility of Flow Measurements in the SMA Using Doppler Ultrasound
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: CCP19-3306-DUS
Record Dates: First submitted 2019-05-06; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Doppler Ultrasound will be performed in all subjects.
  Interventions: Other: Doppler Ultrasound

INTERVENTIONS:
Other: Doppler Ultrasound — Flow measurements using Doppler ultrasound

SUMMARY:
This will be a single center, methodological study in healthy male subjects to evaluate the intra-period, inter-period and inter-observer reproducibility of flow measurements in the superior mesenteric artery, using Doppler Ultrasound.

DETAILED DESCRIPTION:
This will be a single center, methodological study in healthy male subjects, aged 18-50, to evaluate the intra-period, inter-period and inter-observer reproducibility of flow measurements in the superior mesenteric artery, using Doppler Ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male ≥18 and ≤ 50 years of age.
* Subject is a non-smoker for at least 6 months prior to study start.
* Subject has a body mass index between 18-28 kg/m2.
* Subject is judged to be in good health on the basis of medical history and vital signs.
* Subject understands the procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

* Subject has a history of any illness which, in the investigator's opinion, might confound the results of the study.
* Subject has burns, scars, flaps or grafts on the abdomen which, in the investigator's opinion, may interfere with the study assessments.
* Subject has an anatomical anomaly of the SMA as evaluated with DUS during screening which, in the investigator's opinion, may interfere with the study assessments.
* Subject currently uses any prescription or non-prescription drugs on a regular basis which, in the investigator's opinion, might confound the results of the study. Subject has taken 7 days prior to the start of the study any prescription or non-prescription drugs which, in the investigator's opinion, might confound the results of the study.
* Subject is unable to refrain from drinking alcohol 24 hours prior to each study visit or has a history of drug (including alcohol) abuse.
* Subject is unable to refrain from drinking caffeinated beverages (e.g. coffee, tea, cola, …) 24 hours prior to each study visit. Subject is unable to limit their intake of caffeinated beverages to ≤4 cups a day throughout the study.
* Subject has any of the following vital sign measurements at screening: Heart Rate <40 or >100 beats/min, Diastolic Blood Pressure <50 or >90 mmHg, Systolic Blood Pressure <90 or >140 mmHg.
* Subject has been involved in testing an investigational drug in another clinical study within the last 4 weeks.
* Subject is in a situation or has a condition which, in the opinion of the investigator, may interfere with optimal participation in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male volunteers
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Intra-period reproducibility of flow measurements | Interval of 30 minutes between two measurements during study visit 1
  Reproducibility of flow measurements performed during study visit 1 by the same observer.
Intra-period reproducibility of flow measurements | Interval of 30 minutes between two measurements during study visit 2
  Reproducibility of flow measurements performed during study visit 2 by the same observer.
Inter-period reproducibility of flow measurements | Interval of at least 3 days between both study visits
  Reproducibility (i.e. assessing changes) of flow measurements performed during two separate study visits by the same observer
Inter-observer reproducibility of flow measurements | Interval of 15 minutes between two measurements during study visit1
  Reproducibility of flow measurements performed during study visit 1 by two different observers.
Inter-observer reproducibility of flow measurements | Interval of 15 minutes between two measurements during study visit 2
  Reproducibility of flow measurements performed during study visit 2 by two different observers.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Pharmacology, Leuven, Vlaams Brabant, Belgium